CLINICAL TRIAL: NCT06711926
Title: Influence of School Beverage Choice on Hydration Status Cognition and Learning in Primary School Aged Children
Brief Title: Influence of Beverage Choice on Hydration Status Cognition and Learning in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Principal Investigator, Catrin Roberts, PhD, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NorthumbriaU(CR/PR)
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Dehydration in Children; Thirst; Beverage Hydration Index
Keywords: Appetite; Cognition; Gastric emptying
MeSH Terms: interventions — Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Randomised, crossover study.
Who Masked: Participant
Masking Description: Test beverages were presented to the participant in a dark bottle, and were not told which beverage they were consuming for each trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Beverage 1 (Experimental): Distilled water
  Interventions: Other: Distilled water
- Experimental: Beverage 2 (Experimental): Semi skimmed milk
  Interventions: Other: Semi-skimmed milk
- Experimental: Beverage 3 (Experimental): Whey permeate
  Interventions: Other: Whey permeate

INTERVENTIONS:
Other: Distilled water — Participants will receive 600ml distilled water with a strawberry flavour, in four equal aliquots across 30 minutes (150ml every 7.5minutes)
  Arms: Experimental: Beverage 1
Other: Semi-skimmed milk — Participants will receive ~600ml semi-skimmed milk with a strawberry flavour in four equal aliquots across 30minutes (150ml every 7.5minutes).
  Arms: Experimental: Beverage 2
Other: Whey permeate — Participants will receive ~600ml whey permeate (30g sachet, rehydrated with distilled water)with strawberry flavour in four equal aliquots across 30minutes (150ml every 7.5minutes).
  Arms: Experimental: Beverage 3

SUMMARY:
The main aim of this clinical trial is to compare the beverage hydration index of three different beverages in primary school-aged children.The Beverage Hydration Index (BHI), compares the hydration value of beverages against plain water. This study will explore the fluid retention capabilities of semi-skimmed milk, milk permeate, and water.

This study will also investigate:

* Identify the most effective beverage for hydration and the potential cognitive and mood benefits.
* To test if these beverages have any effect on gastric emptying
* To test if these beverages have any effect on appetite.
* To test the acceptability and palpability of semi-skimmed milk, milk permeate, and water in primary school-aged children.

Participants will:

* Take part in three study days (one for each beverage)
* Study day will take part between 9:00AM-12:30PM
* Participants will also record their food and fluid consumption the day before and consume a standardised breakfast before each trial.
* The beverage hydration index will be calculated as the mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
* Blood and urine samples will be taken to measure hydration
* Breath samples will be taken for gastric emptying rate
* COMPASS (Computerised Mental Performance Assessment System), fNIRS (Functional Near Infrared Spectroscopy) and visual analogue scales (VAS) measures will be obtained to assess cognition/mood
* An ad libitum pasta meal will be consumed after the trial to measure appetite, along with blood glucose and GLP-1 and further VAS to measure self reported hunger and fullness.
* A focus group will be held following completion of all three beverage trials, to gather participants opinion of each drink.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 9-11
* Healthy

Exclusion Criteria:

* Psychiatric, neurological or mental disorder.
* Children with any morbidity that might influence hydration status (i.e., renal/cardiovascular/metabolic disease), blood-borne illness, or if they were taking any medications that may impact fluid balance.
* Children that are lactose intolerant
* Children that have any food allergies

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Beverage hydration index | 0 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage hydration index | 60 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage hydration index | 120 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.

SECONDARY OUTCOMES:
Net Fluid Balance | 0 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 60 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total
Net Fluid Balance | 120 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total
Urine Osmolality | -30 minutes before beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 0 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 60 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 120 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Serum osmolality | -30 minutes (before beverage consumption)
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 0 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 30 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 60 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 120 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Gastric emptying rate | -30 minutes (before beverage), 15, 30, 45, 60, 75, 90, 105, 120 minutes (after beverage consumption).
  Test beverages will be infused with 13C-sodium acetate and evaluated using the 13C breath test. Samples will be analysed to determine the ratio of 13CO2 to 12CO2. The change in this ratio from the baseline to post-beverage samples will be expressed as delta over baseline (DOB).
Cognitive function | -45 minutes (before beverage consumption)
  A collection of five cognitive tasks including choice reaction time, simple reaction time, Stroop, Picture recognition and Corsi blocks via Computerised Mental Performance Assessment System (COMPASS)
Cognitive function | 45 minutes (after beverage consumption)
  A collection of five cognitive tasks including choice reaction time, simple reaction time, Stroop, Picture recognition and Corsi blocks via Computerised Mental Performance Assessment System (COMPASS)
Cognitive function | 105 minutes (after beverage consumption)
  A collection of five cognitive tasks including choice reaction time, simple reaction time, Stroop, Picture recognition and Corsi blocks via Computerised Mental Performance Assessment System (COMPASS)
Neuroimaging | -45 minutes (before beverage consumption)
  Functional near-infrared spectroscopy (fNIRS) will monitor changes in the blood oxygenation and blood volume that are related to the human brain function. The headband will be worn whilst participants complete the cognitive tasks.
Neuroimaging | 45 minutes (after beverage consumption)
  Functional near-infrared spectroscopy (fNIRS) will monitor changes in the blood oxygenation and blood volume that are related to the human brain function. The headband will be worn whilst participants complete the cognitive tasks.
Neuroimaging | 105 minutes (after beverage consumption)
  Functional near-infrared spectroscopy (fNIRS) will monitor changes in the blood oxygenation and blood volume that are related to the human brain function. The headband will be worn whilst participants complete the cognitive tasks.
Subjective mood and appetite | -30 minutes (before beverage consumption), 0, 45, 105, 120 and 150minutes (after beverage consumption)
  Mood measured with visual analogue scale (VAS) on 100 mm horizontal lines. Additional VAS will be completed for thirst and appetite. Participants will simply mark a vertical line between the anchored terms, which they feel fittingly, represents how they are feeling at that time. For example, the happiness VAS will have the terms "very happy" printed on the right-hand side of the scale and "very sad" on the left-hand side. The hunger and thirst scales will have 'not hungry or thirsty' printed on the left-hand side and 'very hungry or thirsty' on the right-hand side. A low score will demonstrate that the child had put a mark at the 'not' end of the scale, a high score would show that the child had put a mark at the 'very' end of the scale.
Subjective beverage acceptability | 0 minutes (immediately after beverage consumption)
  Subjective beverage palatability and acceptability measured with visual analogue scale (VAS) on 100 mm horizontal lines. Participants will simply mark a vertical line between the anchored terms, which they feel fittingly, represents how they are feeling at that time. The participants will score terms "sour, sweet, salty, taste, hydrating, stomach bloating, drink again". The score of 0 will indicate they dislike and the score of 100 will indicate they like the beverages.
Ad libitum meal | 120-150 minutes (after beverage consumption)
  Lunchtime food intake will be assessed from a standardised pasta meal offered ad libitum. Energy intake will be calculated based on the amount consumed and the nutritional information provided Nutritics. The meal will be weighed before and immediately after the participant finished eating.
Blood glucose | At 120 minutes and 150 minutes (before after the ad-libitum lunch meal)
  Blood glucose concentrations will be measured instantly using the glucose oxidase method with an automated glucose analyser
Focus group | Following completion of all beverage trials, an average of 8 weeks
  After all participants have completed their trials, a focus group will be held to gather the children's options on the drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Catrin Roberts, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No